CLINICAL TRIAL: NCT04815291
Title: STREAMLoc- Streamlined Localization Using SCOUT® at Biopsy: An Analysis of Process Improvement, Cost Savings and Enhanced Patient Experience.
Brief Title: Streamlined Localization Using SCOUT® at Biopsy (STREAMLoc )
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision.
Sponsor: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCOUT2021
Record Dates: First submitted 2021-03-16; First posted 2021-03-25 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Device (Experimental): Receives SCOUT at biopsy
  Interventions: Device: Receives SCOUT at biopsy

INTERVENTIONS:
Device: Receives SCOUT at biopsy — SCOUT Reflector

SUMMARY:
This registry is intended to demonstrate the utility of SCOUT® in the Canadian public and US healthcare systems with fixed resources and a conservative approach to patient and clinician exposure to harm. The efficacy and safety of this system will be further assessed, as well as the acceptance of clinicians and patients.

DETAILED DESCRIPTION:
This registry is intended to demonstrate the utility of SCOUT® in the Canadian public and US healthcare systems with fixed resources and a conservative approach to patient and clinician exposure to harm (i.e., radiation, COVID-19 exposure, patient emotional trauma). By assessing the utility of reflector insertion at the time of biopsy, this study will be able to measure the impact on patient visits to the breast center for invasive procedures between biopsy and surgery, and quantify this value to the public healthcare system. The efficacy and safety of this system will be further assessed, as well as the acceptance of clinicians and patients.

ELIGIBILITY:
Inclusion Criteria:

1. Woman >18 years and < 80 years of age;
2. Classified as Breast Imaging Reporting and Data System (BI-RADS) 4C or 5;
3. Lesion depth is < 6 cm from skin surface;
4. Non-palpable lesions;
5. Informed consent obtained.

Exclusion Criteria:

1. Multicentric breast cancer;
2. Pregnant or lactating;
3. Known or suspected nickel-titanium allergy.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C Desbiens, MD, Principal Investigator — St. Sacrement
Locations (2):
- Canada (2):
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - St. Sacrement, Québec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Device
Started | 93
Completed | 85
Not Completed | 8
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 4
Not completed — Surgery not planned and subject not operated. | 3

BASELINE CHARACTERISTICS:
Population: Although 93 subjects were enrolled as the overall number of baseline participants, there was one participant that did not have available data.
Arm/Group | Device
Number analyzed (Participants) | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 92

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Invasive Visits
Description: Number of visits to the breast centre for an invasive procedure between biopsy and surgery
Time Frame: through study completion, an average of 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 85
Participants | 5

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Device-related adverse event rate
Time Frame: through study completion; an average of 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 93
Participants | 1

3. Secondary Outcome: Performance
Description: Successful Procedure is absence of close margins (<2mm), positive margins (tumor on ink) or requirement for re-excision.
Time Frame: through study completion; an average of 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 85
Participants | 84

ADVERSE EVENTS:
Time Frame: Adverse events were collected through study completion; average of 6 months.
Description: The following adverse events of interest and device deficiencies were collected: Adverse reaction to material, Device Migration, Inaccurate location detection, Inaccurate deployment, Infection Tissue/vascular trauma, and any AE that, in the opinion of the investigator, has a causal relationship (probable or definite) to the device or procedure, or any device deficiency, whether or not associated with an adverse event. All AEs collected were treatment related.
Arm/Group | Device
All-Cause Mortality (participants affected / at risk) | 0/93
Serious Adverse Events (participants affected / at risk) | 0/93
Other Adverse Events (participants affected / at risk) | 1/93
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device (N=93)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/91/NCT04815291/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT04815291/SAP_001.pdf